CLINICAL TRIAL: NCT01286077
Title: A Phase 2, Multicentre, Randomised, Open-Label, Parallel Group Study to Evaluate the Effect of VELCADE on Myeloma Related Bone Disease
Brief Title: Velcade Consolidation Bone Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR016270; 26866138MMY2060 (Other: Janssen-Cilag International NV); 2008-004264-39 (EudraCT Number)
Record Dates: First submitted 2011-01-27; First posted 2011-01-31 (Estimated); Results first posted 2013-12-30 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-04

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; bortezomib; hematology; bone marrow cancer; Myeloma-related bone disease; bone mineral density; bone markers
MeSH Terms: conditions — Multiple Myeloma; Bone Marrow Neoplasms | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- bortezomib (Experimental): bortezomib (Velcade) 1.6 mg/m² bolus injection on Days 1, 8, 15 and 22 every 5 weeks for 4 cycles
  Interventions: Drug: bortezomib
- Non-treated control (No Intervention): no treatment, observation only

INTERVENTIONS:
Drug: bortezomib — Each cycle will consist of 5 weeks treatment. Subjects in the treatment group will receive: Velcade® 1.6 mg/m2 as an intravenous bolus injection on Days 1, 8, 15, and 22 of each cycle followed by a 13-day rest period (Days 23 to 35) Cycle will be repeated on Day 36. Subjects in the treatment group will receive up to 4 treatment cycles, unless they experience either unacceptable toxicity or if the subject requests to withdraw from the study.
  Arms: bortezomib

SUMMARY:
The purpose of this study is to assess the effect of bortezomib on myeloma-related bone disease, analyzing bone mineral density (BMD) in patients with Multiple Myeloma (MMY) who have received high dose chemotherapy and autologous stem cell transplantation for primary treatment of MMY (single- or double-transplant). Eligible patients will be randomized (study treatment assigned by chance like flipping a coin) to either bortezomib or observation alone. Patients in the bortezomib arm will receive treatment of bortezomib for a total of 4 cycles. All subjects will be followed for a total of 24 months after randomization.

DETAILED DESCRIPTION:
This is a randomized, open-label (all people involved know the identity of the intervention), multicenter, multi-country parallel group study (each group of patients will be treated at the same time) in patients with Multiple Myeloma (MMY) who have received high dose chemotherapy and autologous stem cell transplantation for primary treatment of MMY (single- or double-transplant). The purpose of the study is to assess the effect of bortezomib on myeloma-related bone disease by analyzing bone mineral density. Approximately 80% of patients with MMY may experience myeloma-related bone disease. Myeloma-related bone disease may cause skeletal complications, including bone pain, bone lesions, abnormal fractures and super-elevated calcium concentrations in the blood. This study is investigating the safety and efficacy of an experimental drug, bortezomib, to consolidate the response to the primary treatment compared to no such consolidation treatment. The analyses in this study will be exploratory in nature, since the study will not address any pre-defined statements but is designed to generate valid hypotheses on safety and efficacy issues. Bortezomib is currently marketed for the treatment of different types of cancer including MMY. Bortezomib has been shown to promote bone formation and increase the number of bone-regenerating cells in preliminary studies. In the present study, the effect of bortezomib on bone formation will be assessed by dual energy x-ray absorptiometry (DXA) measuring bone mineral density, which is a measure for the quality of the bone structures. Several bone markers will be measured on serum samples. Bone markers are indicators of the bone activity. Patients will be evaluated for eligibility within a 14-day screening period, after providing written informed consent. Eligible patients will then be randomised to either bortezomib or observation alone. Baseline efficacy and safety assessments should be available on Cycle 1 Day 1 prior to administration of study medication. Randomization will be stratified by bisphosphonate treatment (use or not) at baseline and age (65 years or more versus less than 65 years). The treatment period is defined as the time the patient is actively receiving study treatment. Patients in the bortezomib arm will receive treatment of bortezomib for a total of 4 cycles or until start of alternative MMY treatment if earlier. Each cycle will consist of 5 weeks treatment. Subjects in the treatment group will receive bortezomib 1.6 mg/m2 on Days 1, 8, 15, and 22 of each cycle followed by a 13-day rest period (Days 23 to 35). Bisphosphonate therapy can be administered as medically indicated and according to local practice. Patients are to attend study center visits on Days 1, 8, 15, and 22 of each treatment cycle or at Days 1, 36, 71, and 106 in the observation arm and at end of treatment (EOT) Visit. During these visits, different evaluations will be conducted to follow treatment safety: symptom directed physical examination, vital signs and laboratory tests. In addition, at Day 1 of Cycle 3 (prior to dosing) or Day 71 in the observation arm, patients will be assessed for disease progression or relapse by measurements of M-protein in serum and urine. If needed, absence of M-protein in serum and urine will be confirmed by immunofixation. Additional evaluations may be performed to document patient's clinical status and ability to tolerate additional therapy as clinically indicated. All patients will be followed for a total of 24 months since baseline. After end of the treatment phase, there will be a long-term follow-up period with visits at 4, 6, 12 and 18 months after the EOT Visit. In case the patient started alternative MMY treatment before completing the 18 months of follow-up, study assessments will stop, except for QoL assessments, which are to be continued up to 18 months of follow-up, and for a long-term follow-up for survival, which will be collected every 6 months by either a telephone call or a visit to the study site. The follow-up for survival will continue for all patients until the last patient has completed follow-up. In addition to scheduled visits, patients may have additional visits as clinically indicated. Every patient who was randomized should enter the long-term follow-up phase. Assessment of progressive disease (PD) or relapse from complete response (CR) should be performed according to the International Myeloma Working Group (IMWG) 2009 criteria. Changes in serum and urine M-protein (monoclonal paraprotein) levels will be confirmed by immunofixation in patients without measurable serum and urine M-protein levels. Karnofsky performance status will also be assessed. Safety will be assessed by monitoring of adverse events, physical examination (including neurological/peripheral neurological examinations), vital signs measurements and clinical laboratory tests. A total of two exploratory analyses will be performed for the present study: The first analysis (main analysis) will be presented after completion of the EOT Visit (24-weeks data). The second analysis will be the analysis at the end of the study on 18 months follow-up data. Patients in the bortezomib arm will receive treatment of bortezomib 1.6 mg/m² as a bolus infusion on Days 1, 8, 15, and 22 every 5 weeks for a total of 4 cycles

ELIGIBILITY:
Inclusion Criteria:

* Adult Multiple Myeloma patients in partial response or better after high dose chemotherapy and autologous stem cell transplantation
* Patient fulfills defined laboratory requirements within 14 days before enrolment
* If female, is either postmenopausal for more than 24 consecutive months or surgically sterilized or willing to use an acceptable method of birth control for defined period
* If male, agree to use an acceptable barrier method of contraception and to not donate sperm up to 3 months following treatment

Exclusion Criteria:

* Patient received another antimyeloma or experimental therapy following autologous stem cell transplantation
* Patient has a peripheral neuropathy or neuropathic pain of grade 2 or greater intensity as defined by the NCI common terminology criteria of adverse event (NCI CTCAE) version 3.0
* Patient has an uncontrolled or severe cardiovascular disease within 6 months of enrolment
* Patient has any conditions that would compromise his/her well-being or the completion of the study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2009-09; Primary Completion 2012-11 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (21):
- Austria (3):
  - Feldkirch
  - Graz
  - Vienna
- Brno, Czechia
- Vejle, Denmark
- Germany (3):
  - Hamburg
  - Kiel
  - Mÿnchen
- Athens, Greece
- Sweden (2):
  - Huddinge
  - Stockholm
- Turkey (Türkiye) (7):
  - Adana
  - Ankara
  - Antalya
  - Eskişehir
  - Gebse
  - Istanbul
  - Izmir
- United Kingdom (3):
  - Edinburgh
  - Sheffield Yorks
  - Wakefield

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bortezomib | Non-treated Control
Started | 51 (One patient did not start treatment and was excluded from the Intent to Treat (ITT) population.) | 53 (One patient did not have any post-baseline assessment and was excluded from the ITT population.)
Completed | 41 | 46
Not Completed | 10 | 7
Not completed — Adverse Event | 2 | 0
Not completed — Death | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Intercurrent illness | 1 | 0
Not completed — Non-compliance | 1 | 0
Not completed — The subject starts with alternative MMY | 0 | 3
Not completed — Patient's decision to stop treatment | 3 | 0
Not completed — Progression of disease | 0 | 1
Not completed — refill medication not received in time | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bortezomib | Non-treated Control | Total
Number analyzed (Participants) | 51 | 53 | 104
Age, Continuous [Mean (Full Range); unit: years] | 56.7 [27 to 75] | 54.7 [35 to 73] | 55.7 [27 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 22 | 40
  Male | 33 | 31 | 64

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Bone Mineral Density (BMD) in the Spine at End of Treatment (EOT)
Description: Change from baseline in bone mineral density (BMD) will be assessed by dual energy x-ray absorptiometry scans at baseline and the EOT visit
Time Frame: at screening (i.e. between 14 and 1 days prior to start of treatment) and at end of treatment (EOT), i.e. 24 weeks after randomization or until start of alternative MMY therapy, if earlier
Population: ITT analysis:13 patients in the bortezomib group and 14 patients in the non-treated control group did not have values at the 2 timepoints to allow calculation of the parameter
Measure: Mean (Standard Deviation); unit: g/mm2
Arm/Group | Bortezomib | Non-treated Control
Number analyzed (Participants) | 38 | 39
g/mm2 | 0.0214 (0.0306) | 0.0167 (0.0301)

2. Primary Outcome: Change From Baseline in Bone Mineral Density (BMD) in the Femur at End of Treatment
Description: Change from baseline in bone mineral density (BMD) will be assessed by dual energy x-ray absorptiometry scans at baseline and the end of treatment EOT visit
Time Frame: as for outcome 1
Population: ITT analysis:8 patients in the bortezomib group and 8 patients in the non-treated control group did not have values at the 2 timepoints to allow calculation of the parameter
Measure: Mean (Standard Deviation); unit: g/mm2
Arm/Group | Bortezomib | Non-treated Control
Number analyzed (Participants) | 43 | 45
g/mm2
  Femur neck | 0.0053 (0.0221) | 0.0044 (0.0299)
  Femur total | 0.0071 (0.0151) | 0.0138 (0.0288)

3. Secondary Outcome: Progression Free Survival
Description: The Progression-Free Survival (PFS) was assessed as median number of months from baseline until the first documented sign of disease progression (increase in disease; radiographic, clinical, or both) or death due to any cause, whichever occurred earlier.
Time Frame: Baseline up to end of study (approximately 4 years 7 months)
Population: Full Analysis Set (FAS) included all the randomized subjects who were eligible for efficacy analysis, that is, excluding subjects who did not have baseline and/or post-baseline data.
Measure: Mean (Standard Error); unit: Months
Arm/Group | Bortezomib | Non-treated Control
Number analyzed (Participants) | 46 | 47
Months | 39.56 (2.02) | 31.66 (1.81)

4. Secondary Outcome: Change From Baseline in Biochemical Bone Markers:Carboxyterminal Telopeptide of Type I Collagen (ICTP), Osteocalcin, Bone-specific Alkaline Phosphatase (BAP)
Description: Bone markers (carboxyterminal telopeptide of type I collagen (ICTP), osteocalcin (Oc) and bone-specific alkaline phosphatase (BAP) was measured on serum samples.
Time Frame: Baseline up to end of study (approximately 4 years 7 months)
Population: FAS was used for analysis. "N" (number of subjects analyzed) signifies the subjects evaluable this measure and n=number pf participants analysed for this outcome measure at specific time point. Missing data was imputed by last observation carried forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: Microgram per liter
Arm/Group | Bortezomib | Non-treated Control
Number analyzed (Participants) | 46 | 47
Microgram per liter
  ICTP (n= 44, 42) | -4.11 (4.36) | -3.51 (3.81)
  Osteocalcin (44, 42) | 20.15 (28.79) | 14.59 (5.57)
  BAP (42, 40) | -0.48 (6.08) | -2.11 (4.80)

5. Secondary Outcome: Change From Baseline in Biochemical Bone Markers: Carboxyterminal Collagen Crosslinks (CTX-I)
Description: Change from Baseline in Biochemical Bone Markers: CTX-I was assessed
Time Frame: Baseline up to end of study (approximately 4 years 7 months)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Nanogram per liter
Arm/Group | Bortezomib | Non-treated Control
Number analyzed (Participants) | 42 | 40
Nanogram per liter | -66.50 (258.26) | -77.68 (158.23)

6. Secondary Outcome: Change From Baseline in Biochemical Bone Markers: Dickkopf Homolog 1 (DKK-1)
Description: Bone markers Dickkopf homolog 1 (DKK-1) was measured on serum samples.
Time Frame: Baseline up to end of study (approximately 4 years 7 months)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Picomole per liter
Arm/Group | Bortezomib | Non-treated Control
Number analyzed (Participants) | 43 | 40
Picomole per liter | -39.31 (82.87) | -25.15 (87.20)

7. Secondary Outcome: Number of Patients With Skeletal Events
Description: Number of patients with skeletal-related events (i.e. pathological fracture (vertebral, non-vertebral, combined), radiotherapy, spinal cord compression, orthopaedic surgery, hypercalcaemia) occurring over 24 months study period
Time Frame: Baseline up to end of study (approximately 4 years 7 months)
Population: FAS included all the randomized subjects who were eligible for efficacy analysis, that is, excluding subjects who did not have baseline and/or post-baseline data. "N" (number of subjects analyzed) signifies the subjects evaluable this measure.
Measure: Number; unit: patients
Arm/Group | Bortezomib | Non-treated Control
Number analyzed (Participants) | 42 | 40
patients | 0 | 0

8. Secondary Outcome: Appearance of New Bone Lesions Compared to Baseline
Description: Appearance of new bone lesions assessed by skeletal survey compared to baseline
Time Frame: Baseline up to end of study (approximately 4 years 7 months)
Population: Data could not be summarised statistically due to insufficient data at End of treatment.
Measure: Number; unit: subjects
Arm/Group | Bortezomib | Non-treated Control
Number analyzed (Participants) | 46 | 47
subjects | 0 | 0

9. Secondary Outcome: Change From Baseline in Spine T-score
Description: T score is used to calculate bone mineral density (calcium and other types of minerals) in an area of the bone. T score is the number of standard deviations above or below the mean for a healthy 30 year old adult of the same sex and ethnicity as a participant. This score is calculated from participant's age, gender and race and skeletal site. T score has a mean of '50' and a standard deviation of '10'. T score lower than its mean indicate low bone mineral density.
Time Frame: Baseline up to end of study (approximately 4 years 7 months)
Population: FAS included all the randomized subjects who were eligible for efficacy analysis, that is, excluding subjects who did not have baseline and/or post-baseline data. "N" (number of subjects analyzed) signifies the subjects evaluable this measure. Missing data was imputed by last observation carried forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Bortezomib | Non-treated Control
Number analyzed (Participants) | 13 | 21
T score | 1.2028 (0.2004) | 1.1811 (0.1689)

10. Secondary Outcome: Karnofsky Performance Status
Description: The Karnofsky performance status is a way to quantify cancer patients' general well-being and activities of daily life and runs from 100 to 0, where 100 is "perfect" health and 0 is death.
Time Frame: Baseline up to end of study (approximately 4 years 7 months)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bortezomib | Non-treated Control
Number analyzed (Participants) | 46 | 47
Units on a scale
  Screening | 92.4 (9.2) | 91.7 (7.0)
  Follow-up | 0.0 (11.4) | 0.4 (7.5)

11. Secondary Outcome: Overall Survival
Description: Overall survival defined as time from first treatment of MMY, i.e. day of first dose of induction therapy for MMY to date of death
Time Frame: Baseline up to end of study (approximately 4 years 7 months)
Population: as for outcome 7
Measure: Median (Standard Error); unit: Months
Arm/Group | Bortezomib | Non-treated Control
Number analyzed (Participants) | 46 | 47
Months | 49.90 (1.48) | 47.26 (1.26)

12. Secondary Outcome: Change From Baseline in Quality of Life Assessed by Euro Quality of Life (EQ-5D)
Description: Subjects were asked to rate their general state of health on a Visual analog scale (in millimeter [mm]) ranging from 0 (worst state of health) to 100 (best conceivable state of health) mm.
Time Frame: Baseline up to end of study (approximately 4 years 7 months)
Population: FAS included all the randomized subjects who were eligible for efficacy analysis, that is, excluding subjects who did not have baseline and/or post-baseline data. Missing data was imputed by last observation carried forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Bortezomib | Non-treated Control
Number analyzed (Participants) | 46 | 47
millimeter (mm) | -0.3 (18.4) | 2.9 (22.6)

13. Secondary Outcome: Tumor Response: Percentage of Participants With Very Good Partial Response (VGPR) or Stringent Complete Response (sCR) or Complete Response (CR) Based on International Myeloma Working Group (IMWG) Response Criteria
Description: Tumor response was assessed as VGPR based on IMWG response criteria if, a) serum/urine M protein detectable by immunofixation but not on electrophoresis or; b) greater than or equal to 90% reduction in serum M protein plus urine M protein level less than 100 milligram/24 hour. CR=normal free light chain (FLC) ratio and absence of phenotypically aberrant plasma cells (PC) in bone marrow with a minimum of 3000 total PC analyzed by multiparametric flow cytometry; Complete response (CR) negative immunofixation on the serum and urine and, disappearance of any soft tissue plasmocytomas and <5% plasma cells in bone marrow.
Time Frame: Baseline up to end of study (approximately 4 years 7 months)
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Bortezomib | Non-treated Control
Number analyzed (Participants) | 46 | 47
Percentage of participants | 82.6 (1.48) | 72.3 (1.26)

14. Secondary Outcome: Tumor Response: Percentage of Participants With Stable Disease (SD) or Progressive Disease (PD) Based on International Myeloma Working Group (IMWG) Response Criteria
Description: Tumor response was assessed as SD based on IMWG response criteria as not meeting criteria for CR, VGPR, PR, or progressive disease; PD as Increase of >=25% from lowest response level in any one or more of the following: serum M protein (absolute increase >=0.5 g/dl)c or urine M protein (absolute increase >=200 mg/24 h); or serum/urine M protein unmeasurable: difference between involved and uninvolved free light chain (FLC) levels; absolute increase >10 mg/dL; or % bone marrow plasma cells: absolute value >=10% or definite development of new bone lesions or soft tissue plasmocytomas or definite increase in the size of existing bone lesions or soft tissue plasmocytomas; or development of hypercalcemia attributed solely to the plasma cell proliferative disorder.
Time Frame: Baseline up to end of study (approximately 4 years 7 months)
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Bortezomib | Non-treated Control
Number analyzed (Participants) | 46 | 47
Percentage of participants | 6.5 (1.48) | 19.1 (1.26)

15. Secondary Outcome: Tumor Response: Percentage of Participants With Partial Response (PR) Based on International Myeloma Working Group (IMWG) Response Criteria
Description: Tumor response was assessed as PR based on IMWG response criteria as >=50% reduction of serum and reduction in 24-h urinary M protein by >=90% or to <200 mg/24 h; or serum/urine M protein unmeasurable:>=50% decrease in the difference between involved and uninvolved FLC levels; or serum/urine M protein and FLC assay unmeasurable: >=50% reduction in plasma cells provided baseline bone marrow plasma cell percentage was >=30%; or plus if present at baseline: >=50% reduction in size of soft tissue plasmocytomas.
Time Frame: Baseline up to end of study (approximately 4 years 7 months)
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Bortezomib | Non-treated Control
Number analyzed (Participants) | 46 | 47
Percentage of participants | 8.7 (1.48) | 8.5 (1.26)

ADVERSE EVENTS:
Time Frame: from the time a signed and dated informed consent form is obtained until EOT Visit (24 weeks after randomization) or until the start of subsequent systemic antimyeloma therapy, if earlier
Arm/Group | Bortezomib | Non-treated Control
Serious Adverse Events (participants affected / at risk) | 6/51 | 3/53
Other Adverse Events (participants affected / at risk) | 47/51 | 35/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib (N=51) | Non-treated Control (N=53)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib (N=51) | Non-treated Control (N=53)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 6 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 19 | 0
Dry mouth (Gastrointestinal disorders) | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 4 | 1
Nausea (Gastrointestinal disorders) | 9 | 0
Vomiting (Gastrointestinal disorders) | 8 | 0
Fatigue (General disorders) | 7 | 1
Pyrexia (General disorders) | 8 | 2
Herpes zoster (Infections and infestations) | 4 | 3
Influenza (Infections and infestations) | 1 | 4
Nasopharyngitis (Infections and infestations) | 6 | 4
Upper respiratory tract infection (Infections and infestations) | 9 | 9
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1
Headache (Nervous system disorders) | 3 | 1
Neuralgia (Nervous system disorders) | 5 | 0
Neuropathy peripheral (Nervous system disorders) | 4 | 1
Paraesthesia (Nervous system disorders) | 4 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 10 | 2
Insomnia (Psychiatric disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Rash (Skin and subcutaneous tissue disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the Sponsor for review at least 60 days prior to submission for publication or presentation. No paper that incorporates Confidential Information will be submitted for publication without Sponsor's prior written consent. If requested in writing, such publication will be withheld for up to an additional 60 calendar days. A publication from the individual Study site data will not be published until the combined results have been published